CLINICAL TRIAL: NCT05283421
Title: Improving Diagnostic in Cervical Dysplasia: A Randomized Study With Local Estrogen Prior to Colposcopy
Brief Title: Improving Diagnostics in Cervical Dysplasia
Acronym: IDEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1-23-456
Record Dates: First submitted 2022-02-11; First posted 2022-03-17 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Cervical Cancer
Keywords: Colposcopy; Estrogen
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled double blind multicenter study
Who Masked: Care Provider
Masking Description: A randomization code will be made and given to the hospital pharmacy who will be packing and blind the tablets for the study. The study medicine will be sent to the women with the same/equal etiquette. At the gynecological examination, the colposcopist will not know which study arm the woman is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active estrogen (Active Comparator): Will receive pretreatment with vaginal application of estrogen 30 microgram (three tablets) once a day for 14 days.
  Interventions: Diagnostic Test: Estrogen
- Placebo (Placebo Comparator): Will receive pretreatment with vaginal application with no estrogen (three tablets) once a day for 14 days.
  Interventions: Diagnostic Test: Placebo

INTERVENTIONS:
Diagnostic Test: Estrogen — Women will receive active estrogen treatment or placebo prior to the colposcopic examination
  Other Names: Vagifem
  Arms: Active estrogen
Diagnostic Test: Placebo — Women will receive active estrogen treatment or placebo prior to the colposcopic examination
  Arms: Placebo

SUMMARY:
Cervical cancer is the fourth most common cancer in women worldwide. It is caused by an infection with human papillomavirus (HPV). A persistent infection with HPV is associated with increased risk of precancerous lesions, which may further develop into cervical cancer. To reduce the disease burden, accurate and timely diagnosis of cervical precancerous lesions are crucial.

To identify cervical precancerous lesions, women are referred to colposcopy, which is the most important diagnostic tools to detect cervical precancerous lesions. It allows close visualization of the cervix in order to collect biopsies in the area called transformation zone (TZ), which is where precancerous lesions develop. It is essential for the physician to identify the TZ during colposcopy in order to obtain correct diagnosis. For women aged ≥50 this is often a challenge as TZ naturally with age, will retract further into the cervical canal, making the area for sampling invisible, and thereby the colposcopy inadequate.

Consequently, this increases the risk of developing cancer due to diagnostic delay, and the risk of several colposcopy examinations or overtreatment (cone biopsy), before a final diagnosis is achieved.

Few studies suggest that pretreatment with local vaginal estrogen prior to colposcopy may improve visualization of the TZ. Thereby, obtaining more accurate biopsies from the cervix, and thus making a more accurate and timely diagnosis in the first outpatient visit.

The primary purpose of this study is to evaluate pre-diagnostic treatment with estrogen to improve the diagnosis of women with cervical precancerous lesions, in order to prevent cervical cancer.

The study ia s randomized controlled double-blind multicenter study. The investigators will use information from Danish National Patient registry, and data from the Danish Pathology Data Bank. Enrollment will take place at the Departments of Gynecology in Denmark. Eligible women aged ≥ 50 years will be randomized 1:1 to receive local vaginal estrogen or placebo prior to the colposcopic examination.

The investigators believe the results will provide the prerequisite for obtaining correct diagnosis, and thereby provide basis for choosing the right individualized examination- and treatment plan. The results will also contribute with important knowledge, that may help reduce the incidence and mortality rate of cervical cancer.

DETAILED DESCRIPTION:
Cervical cancer is the fourth most common cancer in women worldwide, and comprises approximately 7% of all new cancers in women. To reduce the disease burden, accurate and timely diagnosis of cervical precancerous lesions are crucial.

Aim:

The aim of this study is to evaluate whether optimizing present procedures can improve diagnosis of precancerous cervical lesions.

The study aims to:

1. Initiate a double blind study to investigate, if the diagnosis of cervical precancerous lesions can be improved among elderly women aged ≥ 50 years, by providing pretreatment with vaginal estrogen prior to the colposcopic examination.

Background:

In Denmark, about 400 women are diagnosed with cervical cancer annually, and around 15.000 women are diagnosed and treated with cervical precancerous lesions. Cervical cancer is preventable through HPV vaccination and screening, yet the incidence rates have stagnated. Cervical cancer is caused by an infection with a high-risk human papillomavirus (HPV), which is a common sexually transmitted disease, with a life-time risk of >80%. In 10-15% of the infected women, the infection becomes persistent, and may cause precancerous lesions (Cervical Intraepithelial Neoplasia, CIN). CIN is graded according to severity (CIN1, CIN2, and CIN3), and can progress and develop into cancer if left untreated. The classification of CIN dictates the treatment course, and surgical treatment (cone biopsy) is recommended in most cases of CIN2 or worse (CIN2+). To identify precancerous lesions, all 23-64-year-old women in Denmark are invited for screening with a cervical cytology sample or an HPV test every third or five years. The cervical cytology sample is classified as mild (low-grade squamous intraepithelial lesion, LSIL) or moderate to severe (high-grade squamous intraepithelial lesion, HSIL). ASCUS is a term used to describe atypical cervical squamous cells of undetermined significance. An abnormal screening sample results in a referral for further examination by colposcopy. It allows close visualization of the cervix in order to detect suspicious lesions, and collection of cervical biopsies.

Diagnostic of cervical precancerous lesions:

Colposcopy is the most important diagnostic tools to detect cervical precancerous lesions and thereby prevention of cervical cancer. The area on the cervix where precancerous lesions and cancer develops is called the transformation zone (TZ), and the squamocolumnar junction (SCJ) refers to the internal margin of the TZ. The TZ is classified as type 1, 2 or 3 according to the visibility of all or part of the upper limit of the SCJ, that is either found completely visible (TZ1), partly visible (TZ2) or not visible (TZ3). To perform optimal examination and obtain a correct diagnosis, it is essential for the physician to identify the TZ. However, the colposcopy procedure may be challenging and performs poorly, especially among elderly women due to natural age-related changes of the cervix. After menopause, the TZ will retract into the cervical canal, which makes visualization of the SCJ and TZ difficult, rendering the colposcopy examination inadequate. Previous studies revealed inadequate colposcopy in up to 30-97%, increasing with age. Consequently, this increases the risk of developing cancer due to diagnostic delay, but also the risk of undergoing several colposcopy examinations or overtreatment by a cone biopsy (thereby also the risks related to surgery), causing adverse psychological outcomes, before a final diagnosis is achieved. Evidence-based practice is lacking on how, especially elderly women should be examined and followed-up in case of inadequate colposcopic examinations. This is a noteworthy public health concern, as elderly women are more likely to be diagnosed with advanced cervical cancer with higher mortality, due to late prognosis and faster disease progression. Furthermore, this group of elderly women is expected to increase in the future, due to the increasing female life expectancy, and due to the extensions of the cervical cancer screening programs in some countries, including Denmark.

Optimizing the colposcopic performance:

A few studies with limited sample sizes (ranging between 35 to 50 participants) suggested that pretreatment with estrogen prior to colposcopy may improve visualization of TZ and consequently improve diagnostics in elderly women. However, the quality of the previous studies is far from adequate and comparable. Furthermore, apart from age, there is also no risk factors described (e.g. previous dysplasia) with respect to the type of TZ as 1, 2 or 3.

Hypotheses for this study:

• Treatment with vaginal estrogen prior to colposcopy will improve the colposcopy performance in women aged ≥ 50 years as compared to standard procedure which is no treatment.

Material and methods:

The study will be designed as a randomized controlled double-blinded multicenter study. Enrollment will be performed at the Departments of Gynecology in Denmark (cities: Randers, Herning, Horsens and Odense). Eligible women will be booked for colposcopy as usual. By using the Danish National Patient registry, the investigators will be able to identify women referred for colposcopy, and collect relevant patient data. This will be combined with data from the nationwide Danish Pathology Data Bank, which will provide the histopathological results of the biopsies. The colposcopic examination will be performed by nurses and physicians who routinely perform colposcopies. Stata version 16 will be used for data analysis, and data will be stored in the RedCap database. A study protocol will be prepared in details. The report of the trial will conform to the CONSORT guidelines, and be reported according to the STARD 2015 guidelines.

Eligible women will be randomized 1:1 prior to examination with either:

A) Pretreatment with vaginal application of estrogen 30 microgram once a day every night for 14 days.

B) Placebo with vaginal application without estrogen once a day every night for 14 days.

Study medication will be mailed to the women after receiving written and telephone informed consent. The colposcopy examination will be performed according to current procedures and the Danish national guidelines (DSOG). All biopsies will be collected in one tube for histopathological evaluation. Patients will after examination be asked to score possible side-effects of the pretreatment.

Statistical consideration:

Assuming that the TZ will be visible in 54% of women aged ≥ 50 years in the group receiving placebo, and 81% in the estrogen pre-treatment group, the investigators will be able to detect an improvement in visibility of TZ of 50% or above. This improvement estimate was based on previous research, and also with reference to a clinically relevant threshold. Thus, with a power of 90% and an alpha value of 5%, a sample size of 62 women in each group will be required. To allow for a protocol violation of 20%, 75 women will be included in each group. After enrollment of approximately 30 women in each group, an inter-rim analysis will be performed.

Feasibility and ethics:

The chosen gynecological departments receive a large number of referrals for this patient group, which will ensure a large enrollment. The study will be reported to the Danish Data Protection Agency, the Central Denmark Region Committee on Biomedical Research Ethics and The Danish Health Authority (Danish Medicine Agency), and also registered as a clinical trial (www.clinicaltrials.gov). The GCP unit will supervise the project. Project information will be given to the women orally and written, and they must understand Danish to accept given information before participation. All information will be anonymized prior to analysis. Participation in the study will not have any consequence for the treatment of the women. The dose of estrogen is within the well-known standard recommendation, with a minimum of side effect. It is widely used and recommended by gynecologists to women aged ≥50 years.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (defined as no bleeding ≥1 year) women referred for colposcopy aged ≥ 50 years.
* Women referred for colposcopy due to a positive HPV test and/or an abnormal cervical cytology.
* Women referred for colposcopy due to previous abnormal cervical histology with minimum 6. months since last colposcopy with biopsies.

Exclusion Criteria:

* Use of estrogen within the last 3 months regardless of administration form.
* previous cervical radiotherapy, cervical amputation and/or cone biopsy
* pregnancy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators evaluate diagnostic for cervical precancerous lesions
Enrollment: 150 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
Scoring of the visibility of the Squamous columnar junction (SCJ) | through study completion, an average of 1 year
  Scoring of the visibility of the SCJ by the colposcopist as visible (TZ1), partly visible (TZ2) or not visible (TZ3) during colposcopic examination.
Number of patients with representation of the transformation zone in the cervical biopsies. | through study completion, an average of 1 year
  Representation of the transformation zone in the cervical biopsies from all patients, evaluating from the pathology registration. When the transformation zone is present, the biopsies have been taken in the correct location of the cervix.

SECONDARY OUTCOMES:
The patients' report on possible side effects during pretreatment through questionnaire | through study completion, an average of 1 year
  The patients' report on possible side effects during pretreatment. Patients will be asked about these experiences through a questionnaire before the examination.
Evaluate the proportion of CIN2+ found in biopsies. | 1 month after the biopsy was collected at colposcopy
  Evaluate the proportion of CIN2+ found in biopsies after pathology analyses
diagnostic conus. | 1 month after the biopsy was collected
  Evaluate the proportion of performed diagnostic conus.
Evaluation of biopsies | 1 month after the biopsy was collected at colposcopy
  explore for each patient which biopsy represent the most severe histopathologic result by comparing the first biopsy with the other three

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Esbjerg, GCP-investigator, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Gynecology and Obstetrics, Randers, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertelsen VM, Tranberg M, Petersen LK, Booth B, Bor P. Improving diagnostic of cervical dysplasia among postmenopausal women aged >/=50 years using local vaginal oestrogen treatment prior to colposcopy: study protocol for a multicentre randomised controlled trial (the IDEAL study). BMJ Open. 2024 Jun 23;14(6):e082833. doi: 10.1136/bmjopen-2023-082833. PMID 38910002